CLINICAL TRIAL: NCT01974323
Title: A Safety and Efficacy Study to Compare Dapsone Dermal Gel With Vehicle Control in Patients With Acne Vulgaris
Brief Title: Safety and Efficacy Study of Dapsone Gel in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 225678-007; NCT02786745 (obsolete NCT alias)
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapsone Gel (Experimental): Dapsone gel applied topically to the face and to affected areas of the trunk once daily for 12 weeks.
  Interventions: Drug: Dapsone Gel
- Dapsone Gel Vehicle (Placebo Comparator): Dapsone gel vehicle applied topically to the face and to affected areas of the trunk once daily for 12 weeks.
  Interventions: Drug: Dapsone Gel Vehicle

INTERVENTIONS:
Drug: Dapsone Gel — Dapsone gel applied topically to the face and to affected areas of the trunk once daily for 12 weeks.
  Arms: Dapsone Gel
Drug: Dapsone Gel Vehicle — Dapsone gel vehicle applied topically to the face and to affected areas of the trunk once daily for 12 weeks.
  Arms: Dapsone Gel Vehicle

SUMMARY:
This study will assess the safety and efficacy of dapsone gel versus vehicle control in patients with acne vulgaris.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, parallel-group, vehicle-controlled study to assess the safety and efficacy of dapsone 7.5% gel versus vehicle administered topically once daily for 12 weeks in patients with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acne vulgaris
* Willing to avoid excessive or prolonged exposure to ultraviolet light (eg, sunlight, tanning beds) throughout the study

Exclusion Criteria:

* Severe cystic acne, acne conglobata, acne fulminans, or secondary acne
* Use of phototherapy devices (eg, ClearLight™), energy-based devices, adhesive cleansing strips (eg, Pond's®, Biore®), or cosmetic procedures (eg, facials, peeling, comedo extraction) in the past week
* Use of anti-inflammatory medications, salicylic acid; corticosteroids, antibiotics, antibacterials (including benzoyl peroxide-containing products [eg, benzamycin]), retinoids; other topical acne treatments (eg, photodynamic therapy, medicated soaps such as those containing benzoyl peroxide, salicylic acid, sulfur, or sodium sulfacetamide) in the past 2 weeks
* Use of birth control pills strictly for acne control

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2238 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- United States (2):
  - Beverly Hills, California
  - Aventura, Florida
- Windsor, Ontario, Canada

REFERENCES:
- [Derived] Tanghetti E, Harper J, Baldwin H, Kircik L, Bai Z, Alvandi N. Once-Daily Topical Dapsone Gel, 7.5%: Effective for Acne Vulgaris Regardless of Baseline Lesion Count, With Superior Efficacy in Females. J Drugs Dermatol. 2018 Nov 1;17(11):1192-1198. PMID 30500141
- [Derived] Tanghetti E, Harper J, Baldwin H, Kircik L, Bai Z, Alvandi N. Once-Daily Topical Dapsone Gel, 7.5%: Effective for Acne Vulgaris Regardless of Baseline Lesion Count, With Superior Efficacy in Females. J Drugs Dermatol. 2018 Nov 1;17(11):1192-1198. PMID 30500140
- [Derived] Tanghetti E, Harper J, Baldwin H, Kircik L, Bai Z, Alvandi N. Once-Daily Topical Dapsone Gel, 7.5%: Effective for Acne Vulgaris Regardless of Baseline Lesion Count, With Superior Efficacy in Females. J Drugs Dermatol. 2018 Nov 1;17(11):1192-1198. PMID 30500139
- [Derived] Thiboutot DM, Kircik L, McMichael A, Cook-Bolden FE, Tyring SK, Berk DR, Chang-Lin JE, Lin V, Kaoukhov A. Efficacy, Safety, and Dermal Tolerability of Dapsone Gel, 7.5% in Patients with Moderate Acne Vulgaris: A Pooled Analysis of Two Phase 3 Trials. J Clin Aesthet Dermatol. 2016 Oct;9(10):18-27. Epub 2016 Oct 1. PMID 27847545

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Started | 1118 | 1120
Completed | 1026 | 1027
Not Completed | 92 | 93
Not completed — Other Reasons | 25 | 28
Not completed — Protocol Violation | 2 | 2
Not completed — Personal Reasons | 15 | 19
Not completed — Lost to Follow-up | 45 | 40
Not completed — Pregnancy | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle | Total
Number analyzed (Participants) | 1118 | 1120 | 2238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.5 (8.15) | 20.4 (7.38) | 20.4 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 618 | 631 | 1249
  Male | 500 | 489 | 989

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Score of 0 (None) or 1 (Minimal) on the 5-point Global Acne Assessment Score (GAAS)
Description: The Investigator evaluated the patient's acne severity using the 5-point GAAS scale with 0 being none and 4 being severe. The complete scale is as follow: Grade 0 (none) = No evidence of facila acne vulgaris; Grade 1 (minimal) = Few noninflammatory lesions (comedones) are present, a few inflammatory lesions (papules/pustules) may be present, no nodulo-cyctic lesions are allowed; Grade 2 (mild) = Several to many noninflammatory lesions (comedones) are present, a few inflammatory lesions (papules/pustules) are present, no nodulo-cystic lesions are allowed; Grade 3 (moderate) = Many noninflammatory (comedones) and inflammatory lesions (papules/pustules) are present, no nodulo-cystic lesions are allowed; Grade 4 (severe) = Significant degree of inflammatory disease, papules/pustules are a predominant feature, a few nodulo-cystic lesions may be present, comedones may be present.
Time Frame: Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Percentage of Patients | 29.8 | 20.9

2. Primary Outcome: Change From Baseline in Inflammatory Facial Lesion Counts
Description: The Investigator evaluated the patient's inflammatory lesions (papule, pustule and nodule/cyst). A negative change from baseline indicates a reduction in lesion counts (improvement) and a positive change from baseline indicates an increase in lesion counts (worsening).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Error); unit: Number of Inflammatory Lesions
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Number of Inflammatory Lesions
  Baseline | 29.6 (0.23) | 30.0 (0.23)
  Change from Baseline at Week 12 | -15.6 (0.35) | -14.0 (0.35)

3. Primary Outcome: Change From Baseline in Noninflammatory Facial Lesion Counts
Description: The Investigator evaluated the patient's noninflammatory lesions (papule, pustule and nodule/cyst). A negative change from baseline indicates a reduction in lesion counts (improvement) and a positive change from baseline indicates an increase in lesion counts (worsening).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Error); unit: Number of Noninflammatory Lesions
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Number of Noninflammatory Lesions
  Baseline | 46.7 (0.46) | 46.7 (0.46)
  Change from Baseline at Week 12 | -20.8 (0.55) | -18.7 (0.55)

4. Secondary Outcome: Change From Baseline in Total Lesion Counts
Description: The Investigator evaluated the patient's inflammatory (papule, pustule and nodule/cyst) and non-inflammatory (blackhead and whitehead) lesions. A papule is a small, red, solid elevation less than 1.0 cm in diameter, a pustule is a small, circumscribed elevation of the skin that contains yellow-white exudate and a nodule/cyst is a circumscribed, elevated, solid lesion generally more than 0.5 cm in diameter with palpable depth. The total lesion count was the sum of the inflammatory and non-inflammatory lesion counts. A negative change from baseline indicates a reduction in lesion counts (improvement) and a positive change from baseline indicates an increase in lesion counts (worsening).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Least Squares Mean (Standard Error); unit: Total Lesion Counts
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Total Lesion Counts
  Baseline | 76.4 (0.56) | 76.9 (0.56)
  Change from Baseline at Week 12 | -36.2 (0.76) | -32.3 (0.75)

5. Secondary Outcome: Percentage Change From Baseline in Total Lesion Counts
Description: The Investigator evaluated the patient's Inflammatory (papule, pustule and nodule/cyst) and Non-inflammatory (blackhead and whitehead) lesions. A papule is a small, red, solid elevation less than 1.0 cm in diameter, a pustule is a small, circumscribed elevation of the skin that contains yellow-white exudate and a nodule/cyst is a circumscribed, elevated, solid lesion generally more than 0.5 cm in diameter with palpable depth. The total lesion count was the sum of the inflammatory and non-inflammatory lesion counts. A negative percent change from baseline indicates a reduction in lesion counts (improvement) and a positive percent change from baseline indicates an increase in lesion counts (worsening).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Least Squares Mean (Standard Error); unit: Percent Change in Lesion Count
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Percent Change in Lesion Count | -48.9 (0.97) | -43.2 (0.97)

6. Secondary Outcome: Percentage of Patients Reporting "Very Good" or "Excellent" on Item 10 of the 5-Point Acne Symptom Impact Scale (ASIS)
Description: The patient assessed the impact of their acne vulgaris on the look of their face using item 10 on the 5-point ASIS. Item 10 scores range from 1 (Excellent) to 5 (Bad). The percentage of patients who had an ASIS score of 4 (Fair) or 5 (Bad) at baseline and who reported "Very good" or "Excellent" at Week 12 are reported.
Time Frame: Week 12
Population: Intent-to-Treat: all randomized patients with data at this time point
Measure: Number; unit: Percentage of Patients
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 926 | 961
Percentage of Patients | 24.2 | 22.0

7. Secondary Outcome: Change From Baseline in the 9-Item ASIS Sign Domain Score
Description: The patient assessed signs of acne vulgaris using the ASIS. The sign domain is a composite of 9 items of the 17 items on the overall scale. Each of the items is assessed on a 5-point scale: 0 (best) to 4 (worst). The sign domain score is calculated as the average of the 9 items for a total possible score of 0 to 4. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Scores on a Scale
  Baseline | 2.04 (0.627) | 2.07 (0.612)
  Change from Baseline at Week 12 | -0.74 (0.700) | -0.68 (0.675)

8. Secondary Outcome: Percentage of Patients Reporting at Least a 1-Grade Improvement From Baseline in Facial Oiliness on a the 5-Point ASIS Scale
Description: The patient assessed their facial oiliness using item 1 on the 5-point ASIS. Item 1 scores ranged from 0 (Not at all oily) to 4 (Very oily). The percentage of patients who reported at least a 1-grade improvement from baseline in their facial oiliness are reported.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Percentage of Patients | 48.5 | 49.3

9. Secondary Outcome: Percentage of Patients Reporting at Least a 1-Grade Improvement From Baseline in Facial Redness on a the 5-Point ASIS Scale
Description: The patient assessed their facial redness using item 8 on the 5-point ASIS. Item 8 scores ranged from 0 (Not at all red) to 4 (Very red). The percentage of patients who reported at least a 1-grade improvement from baseline in their facial redness are reported.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Number analyzed (Participants) | 1118 | 1120
Percentage of Patients | 53.8 | 52.9

ADVERSE EVENTS:
Description: The Safety Population was used to assess adverse events and serious adverse events. The Safety Population included all patients who were treated with at least 1 application of study treatment
Arm/Group | Dapsone Gel | Dapsone Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 4/1117 | 4/1118
Other Adverse Events (participants affected / at risk) | 0/1117 | 0/1118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dapsone Gel (N=1117) | Dapsone Gel Vehicle (N=1118)
Peritoneal Haematoma (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Helicobacter Infection (Infections and infestations) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/618 | 1/631 — FEMALES ONLY
Alchoholism (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.